CLINICAL TRIAL: NCT06044311
Title: A Window of Opportunity Trial Evaluating the Oral TGF-beta Receptor I Inhibitor Vactosertib in Patients Undergoing Standard of Care Chemoradiotherapy for Locally Advanced Esophageal Adenocarcinoma
Brief Title: Oral TGF-beta Receptor I Inhibitor Vactosertib in SOC Chemoradiotherapy for Esophageal Adenocarcinoma
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Sakti Chakrabarti (Other)
Responsible Party: Sponsor-Investigator, Sakti Chakrabarti, Principal Investigator, Case Comprehensive Cancer Center
Organization: Case Comprehensive Cancer Center (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CASE1223
Record Dates: First submitted 2023-09-07; First posted 2023-09-21 (Actual); Last update posted 2025-02-24 (Actual); Status verified 2025-02

CONDITIONS: Adenocarcinoma Esophagus; Locally Advanced Adenocarcinoma; Siewert Type I Adenocarcinoma of Esophagogastric Junction; Siewert Type II Adenocarcinoma of Esophagogastric Junction
MeSH Terms: conditions — Adenocarcinoma Of Esophagus | interventions — vactosertib; Carboplatin

STUDY DESIGN:
Intervention Model Description: This study is a phase 2, single-arm, Simon two-stage design. 15 participants will be enrolled in the first stage, with the potential of expanding to an additional 10 participants.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Vactosertib + Chemoradiotherapy (Experimental): Vactosertib orally, 200 mg twice daily for five days a week for 2 weeks, followed by standard of care chemoradiotherapy, followed by Vactosertib for 4 weeks after standard of care chemoradiotherapy
  Interventions: Drug: Vactosertib; Drug: Standard of Care Chemotherapy; Radiation: Concurrent Radiation

INTERVENTIONS:
Drug: Vactosertib — 200 mg orally, twice daily for five days a week, for 2 weeks and again for 4 weeks after chemoradiotherapy.
  Other Names: Oral TGF-beta Receptor I Inhibitor
Drug: Standard of Care Chemotherapy — Neoadjuvant chemotherapy treatment as per standard of care.
  Other Names: Carboplatin; Paciltaxel
Radiation: Concurrent Radiation — Neoadjuvant radiation treatment as per standard of care.

SUMMARY:
This interventional clinical trial aims to find ways of improving treatments for individuals with esophageal cancer. Laboratory-based studies show that using medicines that affect a protein called TGF-beta (TGFβ) can kill esophageal cancer cells in individuals who have localized esophageal adenocarcinoma and are being considered for standard-of-care chemoradiation prior to surgery. Participants of this study will take a pill called vactosertib for two weeks before starting standard of care chemoradiation. At the end of the two weeks of taking vactosertib, participants will have a Positron Emission Tomography Computer Assisted Tomography (PET CT) scan and undergo an endoscopy with a biopsy to determine if the vactosertib is working. After chemoradiation, participants will take vactosertib again for four weeks and then be considered for surgery.

DETAILED DESCRIPTION:
Esophageal adenocarcinoma (EAC) is an aggressive malignancy with limited effective treatment options. In localized EAC (clinical stages II and III), the standard of care is pre-operative concurrent chemoradiation (CRT) followed by surgical resection, which results in pathologic complete response (pCR) in approximately 20% of participants, but with high rates of post-operative recurrence. It was recently discovered that EACs are driven by signaling through TGFβ Receptor I (TGFβRI), and in vivo models of EAC show tumor reduction by targeting this pathway with a novel small molecule inhibitor of TGFβRI called vactosertib. In this study, participants who have locally advanced EAC will be treated with vactosertib before and after standard of care chemoradiation to take advantage of natural windows of opportunity during which participants are being planned for their standard of care treatments.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must have histologically or cytologically confirmed poorly differentiated or Grade 3 adenocarcinoma of the esophagus or gastroesophageal junction, clinical Stage II or III who are appropriate for concurrent chemoradiotherapy with carboplatin and paclitaxel or FOLFOX as per standard of care. Clinical staging appropriate:

  * cT2 N0 with high-risk lesions including lymphovascular invasion, tumors ≥ 3cm in size, or poorly differentiated histology, or
  * cT1b-cT2, N+, or
  * cT3-cT4a, any N
* Subjects must be deemed a potential surgical candidate by a thoracic surgeon, surgical oncologist, or surgeon who is qualified to perform an esophagectomy.
* Subjects must NOT have received prior chemotherapy, immunotherapy, or radiation therapy for management of this malignancy (prior ablations or localized therapies for Barrett's metaplasia are acceptable).
* Age ≥18 years. Because no dosing or adverse event data are currently available on the use of vVactosertib in subjects ≤18 years of age, children are excluded from this study.
* ECOG Performance status ≤2
* Subjects must have normal organ and marrow function as defined below:

  * Serum total bilirubin <2 mg/dl. If known Gilbert syndrome, total bilirubin must be <3mg/dl
  * AST (SGOT) ≤ 2.5 X institutional upper limit of normal
  * ALT (SGPT) ≤ 2.5 X institutional upper limit of normal
  * Serum Creatinine ≤ 1.5 X institutional upper limit of normal
  * Hemoglobin ≥ 7.5 g/dL
  * Absolute neutrophil count ≥ 1,500/mcL
  * Platelet count ≥ 100,000/mcL
* Subjects must have no contraindication to receiving recommended concurrent chemotherapy as per standard of care.
* Subjects must have no contraindication to receiving radiation as per standard of care.
* Women of child-bearing potential and sexually active men with female partners of child-bearing potential must agree to abstain from sexual intercourse for the duration of their participation in the study or agree to use highly effective methods of contraception. This is expected for the entire duration of the study period and up to 6 months after the last dose. Highly effective methods of contraception include: female sterilization (tubal ligation, bilateral oophorectomy, and/or hysterectomy); male sterilization (at least 6 months prior to screening); intrauterine device; and oral, injected, or implanted hormonal contraception AND barrier methods of contraception. Women of child-bearing potential must have documented negative pregnancy test prior to start of investigational treatment regimen.
* Subjects must have the ability to understand and the willingness to sign a written informed consent document.
* Subjects must be able to swallow oral medication.
* Subjects must be willing to undergo endoscopic biopsy and PET CT on trial.

Exclusion Criteria:

* Subjects receiving any other investigational agents. Proton-beam radiation is acceptable, if it is considered standard of care in the opinion of the treating radiation oncologist.
* Subjects with active malignancy within the past 3 years, except if locally curable cancers that have been apparently cured such as non-melanoma cutaneous malignancy, superficial bladder cancer, or carcinoma in situ of the breast or cervix.
* History of allergic reactions to carboplatin, paclitaxel or fluorouracil, oxaliplatin, or vactosertib.
* Subjects with contraindication to radiation therapy.
* Subjects with contraindication to carboplatin and paclitaxel or FOLFOX chemotherapy as per standard of care.
* Subjects with uncontrolled intercurrent illness including, but not limited to ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Pregnant or breastfeeding women are excluded from this study because cytotoxic agents and radiation therapy have the potential for teratogenic or abortifacient effects. Because there is an unknown, but potential risk for adverse events in nursing infants secondary to treatment of the mother with chemotherapy, breastfeeding should be discontinued if the mother participates in the trial. These potential risks may also apply to other agents used in this study.
* HIV-positive patients are ineligible because of the potential for pharmacokinetic interactions with chemotherapeutic agents and because of a potential risk of worsening HIV viral load in response to TGFβ signaling inhibition. In addition, these patients are at increased risk of lethal infections when treated with marrow suppressive therapy.
* Chronic active untreated hepatitis B or C infection. (Assessments should include Hepatitis B Surface AB, Hepatitis B Surface AG, Hepatitis B Core AB - Total, Hepatitis B Core AB, IGM, Hepatitis C AB).
* Treated viral hepatitis patients with undetectable viral load are excluded because there is an enhanced risk of reactivation of the virus. Apart from the potential reactivation risk, the hepatitis-induced liver damage may delay or even cause discontinuation of chemotherapy.
* Viral hepatitis patients receiving antiviral therapy are ineligible because of the potential for pharmacokinetic interactions with chemotherapeutic agents.
* Subject who is taking prohibited medications when using vactosertib as following (refer to APPENDIX III). A minimal washout period of 5 half-lives for the following drugs is recommended prior to the first dosing.

  * Concurrent use of drugs or foods that are known strong CYP3A4 inhibitors including but not limited to grapefruit juice, itraconazole, ketoconazole, lopinavir/ritonavir, mibefradil, voriconazole. The topical use of these medications (if applicable), such as 2% ketoconazole cream, may be allowed.
  * Concurrent use of drugs that are known potent CYP3A4 inducers including but not limited to phenytoin, rifampin, St. John's wort.
  * Concurrent use of drugs that are CYP3A4, CYP1A2, CYP2B6 substrates with narrow therapeutic indices including but not limited to theophylline, astemizole, cisapride, cyclosporine, dihydroergotamine, ergotamine, sirolimus, tacrolimus, terfenadine (astemizole, cisapride, and terfenadine have been withdrawn from the US market).
  * Concurrent use of drugs that are sensitive CYP3A4, CYP1A2, CYP2B6 substrates including but not limited to efavirenz, darunavir, dasatinib, everolimus, lopinavir, midazolam, sirolimus, ticagrelor.
* QTc interval ≥470 ms calculated from 12-lead ECG at baseline.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2024-09-30 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-06-01 (Estimated)

PRIMARY OUTCOMES:
Metabolic Response | At two weeks post treatment
  Determine if two-week treatment with single agent vactosertib induces metabolic response by PET CT imaging in primary EAC tumors. This will be measured as the rate of tumors that have decreased FDG tracer uptake by >= 35% SUV on PET CT after 2 week treatment with vactosertib.

SECONDARY OUTCOMES:
Pathological Response | At approximately 14 weeks from starting treatment
  Evaluate the pathological response at the time of surgery after the combination therapy of CRT followed by vactosertib in patients with locally advanced EAC. This will be defined by the rate of pathological complete response at the time of surgical resection.
Correlate baseline expression | At approximately 14 weeks from starting treatment
  Correlate baseline expression of HNF4A with clinical response to vactosertib. HNF4A expression will be measured by immunohistochemistry and positive or negative expression will be correlated with rate of pathological complete response and metabolic response.
Ability to take vactosertib before and after standard of care chemoradiation | At approximately 14 weeks from starting treatment
  Determine if oral vactosertib is feasible in treatment of locally advanced EAC prior to and after CRT. Feasibility will be measured as the rate of patients able to complete >= 75% of planned doses of vactosertib.

CONTACTS AND LOCATIONS:
Overall Officials: Sakti Chakrabarti, MD, Principal Investigator — University Hospitals Cleveland Medical Center, Case Comprehensive Cancer Center
Locations (1):
- University Hospitals Seidman Cancer Center, Case Comprehensive Cancer Center, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Compiled and analyzed patient data will be published upon study completion. Publisher may request Protocol and Statistical Analysis Plan